IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

Cancer research studies are coordinated by physicians and scientists from Cleveland Clinic, University Hospitals and Case Western Reserve University (CWRU) through the NIH National Cancer Institute (NCI) designated Case Comprehensive Cancer Center (Case CCC). The goal of this collaboration is to enhance cancer treatment and research in Northeast Ohio. This study is being offered at Cleveland Clinic (CC) and University Hospitals (UH).

# What is the usual approach to my breast cancer?

The standard approach to the treatment of metastatic triple-negative breast cancer (breast cancer that has spread to other organs) is chemotherapy (drugs given through a vein) with carboplatin and nab-paclitaxel (two specific chemotherapy drugs).

# What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example:

- you may choose to have the usual approach described above
- you may choose to take part in a different study, if one is available
- you may choose comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

# Why is this study being done?

The purpose of this study is to see how effective the combination of the two chemotherapy drugs (carboplatin and nab-paclitaxel) are when added to a third drug, pembrolizumab.

Pembrolizumab is an investigational (experimental) drug that works by stimulating your immune system, allowing it to target and destroy cancer cells. Pembrolizumab is experimental because it is not approved by the Food and Drug Administration (FDA) for this type of breast cancer treatment.

# What are the study groups?

All study participants will get the same study intervention. It will include receiving treatment containing carboplatin, nab-paclitaxel, and pembrolizumab (also referred to as CNP).

For participants who are unable to tolerate all of the drugs being given the study doctor may allow them to continue to receive treatment with pembrolizumab alone.

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

# CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

A total of approximately 30 patients will be enrolled University Hospitals Cleveland Medical Center and Cleveland Clinic.

# How long will I be in this study?

You will receive the CNP for up to 24 months. After you finish CNP, your doctor will see you for safety evaluation after 30 days. Then, you will be followed by phone calls only. This is called long-term follow-up. This long-term follow-up can be completed over the phone with a study nurse. You will be followed every 3 months up to two years, then every 6 months up to 5 years, and then annually for up to ten years.

# What extra tests and procedures will I have if I take part in this study?

Most of the exams, tests, and procedures you will have are part of the usual approach for your cancer. However, there may be an additional biopsy that you will need to have if you take part in this study.

#### Research biopsies

Tumor biopsies will be done to check the characteristics of your tumor. Your tumor has cells that could be affected by the study drug. If your tumor is accessible, a tumor biopsy will be done.

A tumor biopsy is the removal of a small (pencil eraser-sized) circle of tumor using a cookie cutter-like instrument. The duration of the biopsy procedure is approximately 30 minutes. The biopsy instrument will be placed into the tumor by a physician. The procedure will be done using local anesthesia to minimize discomfort from the biopsy. During a biopsy of the breast, you will be asked to lie flat and a doctor will clean the area on your breast. The doctor will then numb the area with a local anesthetic so that you do not feel the biopsy. The doctor will ask you to hold your breath and not move while he or she places the needle into your tumor and withdraws a small core of tissue which remains trapped inside the needle. This tissue sample will then be forwarded to a research laboratory for further studies.

# Before you begin the study:

You will need to have the following exams, tests or procedures to find out if you can be in the study. These exams, tests or procedures are part of regular cancer care and may be done even if you do not join the study. If you have had some of them recently, they may not need to be

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

# **CONSENT FOR CANCER RESEARCH**

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

repeated. This will be up to your study doctor.

- You will need to supply a complete list of your current medications to the study doctor. This includes over-the-counter medications and herbal supplements.
- The study team will ask you questions about your demographics (examples are sex, race, age, etc.) and your medical history
- Physical exam
- Vital signs (including blood pressure, temperature and pulse)
- Height/Weight
- The study team will ask you how you are currently feeling and your ability to do your daily tasks (also called performance status).
- Routine blood tests (serum chemistry and CBC complete blood count)
- A pregnancy test if you are a woman.
- Tests to measure your tumor. This could be any of the following tests:
  - CT a series of detailed pictures of areas inside the body. The pictures are taken from different angles.
  - $\blacksquare$  MRI a procedure in which radio waves and a powerful magnet linked to a computer is used to make detailed pictures of inside the body.
  - Bone Scan a scan to show any new growth or disease in your bones.

# During the study the following will be additional research procedures:

- A tumor biopsy sample will be collected for research purposes and is required for this study. This will be used to study your cancer in relation to the study drugs CNP. This may be an additional biopsy if your previous biopsy was from too long ago.
- After the research biopsy has been completed, you will receive the following drugs:
  - C, Carboplatin, will be administered intravenously (IV, through a vein) on day 1 of each 21-day cycle. Carboplatin administration may take approximately 60 minutes.
  - o N, Nab-paclitaxel, will be administered IV on days 1, 8 and 15 of each 21-day cycle. Nab-paclitaxel administration may take approximately 30 minutes.
  - o P, Pembrolizumab, will be administered IV on day 15 of each 21-day cycle. Pembrolizumab administration may take approximately 30 minutes.
- After you have completed 3 full cycles of CNP, you will undergo repeat tests to measure your tumor with CTs, MRIs and bone scan, as described above. If these tests show that the

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

metastatic tumor is stable or shrinking, your doctor may choose to continue treatment with CNP.

• An additional biopsy may be done if you agree to this research procedure. It is not required to be part of the main study. This is described in detail on page

# What possible risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work or home and spend more time in the hospital or doctor's office than usual
- You may be asked sensitive or private questions which you normally do not discuss

The CNP therapy used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood and will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drug(s)/study approach. Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.

Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.

The tables below show the most common and the most serious side effects that researchers know about. There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

Possible side effects of carboplatin, which is the usual approach for this type of cancer:

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

# **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving **carboplatin** more than 20 and up to 100 may have:

- Pain at place of injection
- Nausea and vomiting
- Unusual tiredness or weakness

# OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **carboplatin** from 4 to 20 may have:

- Black, tarry stools
- Blood in urine or stools
- Cough or hoarseness, accompanied by fever or chills
- Fever or chills
- Lower back or side pain, accompanied by fever or chills
- Numbness or tingling in fingers or toes
- Painful or difficult urination, accompanied by fever or chills
- Pinpoint red spots on skin
- Skin rash or itching
- Unusual bleeding or bruising
- Unusual tiredness or weakness
- Constipation or diarrhea
- Loss of appetite
- Reduced amount of platelets in the blood: may cause bruising, nosebleeds, or bleeding gums

# RARE, AND SERIOUS

In 100 people receiving **carboplatin** 3 or fewer may have:

- Blurred vision
- Ringing in ears
- Sores in mouth and on lips
- Wheezing

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

Possible side effects of **nab-paclitaxel**, which is the usual approach for this type of cancer: **COMMON, SOME MAY BE SERIOUS** 

In 100 people receiving **nab-paclitaxel** more than 20 and up to 100 may have:

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

# Possible side effects of **nab-paclitaxel**, which is the usual approach for this type of cancer: **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving **nab-paclitaxel** more than 20 and up to 100 may have:

- Black or tarry stools
- Blurred vision
- Burning, numbness, tingling, or painful sensations
- Confusion
- Cough or hoarseness with fever or chills
- Dizziness, faintness, or lightheadedness when getting up suddenly from a lying or sitting position
- Feeling of warmth
- Fever or chills
- Lower back or side pain
- Painful or difficult urination
- Pale skin
- Redness of the face, neck, arms, and occasionally, upper chest
- Shortness of breath
- Skin rash or itching
- Sore throat
- Sweating
- Troubled breathing with exertion
- Ulcers, sores, or white spots in the mouth
- Unsteadiness
- Unusual bleeding or bruising
- Unusual tiredness or weakness
- Weakness in the arms, hands, legs, or feet
- Bleeding, blistering, burning, coldness, discoloration of the skin, feeling of pressure, hives, infection, inflammation, itching, lumps, numbness, pain, rash, redness, scarring, soreness, stinging, swelling, tenderness, tingling, ulceration, or warmth at the injection site
- Cracked lips
- Diarrhea
- Difficulty with swallowing
- Hair loss
- Nausea or vomiting
- Numbness, burning, or tingling in the hands or feet

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

Possible side effects of **nab-paclitaxel**, which is the usual approach for this type of cancer: **COMMON, SOME MAY BE SERIOUS** In 100 people receiving **nab-paclitaxel** more than 20 and up to 100 may have: Pain in the joints or muscles, especially in the arms or legs Thinning of the hair

# OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **nab-palitaxel** from 4 to 20 may have:

Blood in the urine or stools

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

# OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **nab-palitaxel** from 4 to 20 may have:

- Difficult or labored breathing
- Pinpoint red spots on the skin
- Shortness of breath (severe)
- Slow heartbeat
- Tightness in the chest
- Wheezing
- Reduced amount of platelets in the blood: may cause bruising, nosebleeds, or bleeding gums

# **Incidents unknown:**

Some people have reported when receiving **nab-paclitaxel**:

- Anxiety
- Blue lips, fingernails, or skin
- Difficult or troubled breathing
- Fainting
- Fast heartbeat
- Irregular, fast or slow, or shallow breathing
- Sudden shortness of breath

In addition to side effects outlined above, you may also experience the possible side effects of **Pembrolizumab** listed below.

Pembrolizumab which is approved in the USA and some other countries is available by prescription to treat several different cancers, but may not be approved to treat your type of cancer.

Pembrolizumab works by helping your immune system fight your cancer.

However, pembrolizumab can also cause your immune system to attack normal organs and tissues in your body and can affect the way they work, which can result in side effects. These side effects may be serious (i.e. causing hospitalization or be life-threatening), may result in

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

death, and/or may occur after you stop taking pembrolizumab. These side effects can affect more than one of your normal organs and tissues at the same time.

#### **VERY COMMON**

Out of 100 people who receive pembrolizumab, 20 or more people may have the following:

- Itching of the skin
- Loose or watery stools
- Cough

# **COMMON**

Out of 100 people who receive pembrolizumab at least 5 but less than 20 people may have:

- Joint pain
- Rash
- Fever
- Back pain
- Pain in your belly
- Loss of skin color
- Not enough thyroid hormone so you may feel tired, gain weight, feel cold, have infrequent or hard stools (hypothyroidism)
- Low levels of salt in the blood that may cause you to feel tired, confused, have a headache, muscle cramps and/or feel sick to your stomach (hyponatremia)

# **UNCOMMON**

Out of 100 people who receive pembrolizumab, at least 1 but less than 5 people may have the following:

- Too much thyroid hormone so you may feel anxious, angry, have trouble sleeping, feel weak, tremble, sweat, feel tired, have loose and watery stools (hyperthyroidism)
- Inflammation of the lungs so you may feel short of breath and cough (pneumonitis)
- Infusion reaction, where you may feel dizzy or faint, flushed, get a rash, have a
  fever, feel short of breath, experience a decrease in your blood pressure at the
  time of receiving your infusion (IV) or just after, or have pain at the site of
  infusion

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

• Inflammation of the bowels/gut which may cause severe pain in your belly with loose or watery stools and black, tarry, sticky stools or stools with blood or mucus (colitis)

Inflammation of the skin so you may have peeling of the skin, itchiness, and/or skin redness. The skin inflammation (i.e. peeling, itching and redness) could also be widespread throughout your body. More severe skin reactions may involve the inside of your mouth, the surface of your eye and genital areas, and/or may cause the top layer of your skin to peel from all over your body which can cause severe infection (Severe skin reactions, including Stevens-Johnson syndrome or toxic epidermal necrolysis)

# RARE, SOME MAY BE SERIOUS

Out of 100 people who receive pembrolizumab, less than 1 person may have the following:

- Inflammation of the liver that may make you feel sick to your stomach and vomit, feel like not eating, feel tired, have a mild fever, a pain in the right side of your belly, yellow eyes and skin, and dark urine (hepatitis)
- Inflammation of the pituitary gland (a gland in the head), which may cause you to feel sick to your stomach or have headaches, changes in your behavior, double vision, few to no menstrual cycles, weakness, vomiting and dizziness or fainting (hypophysitis)
- Adrenal glands (glands on top of the kidneys) that may not make enough hormone which could cause tiredness, weight loss, muscle weakness, feeling faint, having joint, muscle and belly aches, nausea, vomiting, loose or watery stools, fever, salt craving, and sometimes darkening of the skin like a suntan (adrenal insufficiency)
- Inflammation of the kidney so you may pass less urine or have cloudy or bloody urine, swelling and low back pain (nephritis)
- Inflammation of the muscles so you may feel weak or pain in the muscles (myositis)
- Inflammation of the pancreas, (a gland in your abdomen that controls sugar levels) so you may have severe pain in the top part of your belly that may move to the back, feel sick to your stomach, and vomiting that gets worse when you eat (pancreatitis)
- Inflammation of the eye so you may have eye redness, blurred vision, sensitivity to light, eye pain, see floaters or have headaches (uveitis)
- Type 1 Diabetes, a condition that can cause too much sugar in your blood, feeling thirstier than usual, frequent urination and weight loss. You are likely to need regular insulin shots.
- Inflammation of the nerves that may cause pain, weakness or tingling in the hands and feet, and may spread to the legs, arms and upper body leading to severe muscle

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

weakness and possibly temporary paralysis(Guillain-Barré syndrome)Inflammation of the middle layer of your heart wall that may cause your heart to have difficulty pumping blood throughout your body, which can cause chest pain, shortness of breath and swelling of the legs. You may experience a fast or irregular heartbeat that may cause dizziness or fainting (myocarditis)

- Inflammation of the thyroid gland, an organ that makes and stores thyroid hormones. This condition may lead to change in your heart rate, blood pressure, body temperature, and the rate at which food is converted into energy (thyroiditis)
- A condition that may make you feel weak and tired and may cause drooping of the eyelids, blurred or double vision, difficulty swallowing, slurred speech, weakness in your arms and legs, or difficulty breathing (myasthenic syndrome/myasthenia gravis including exacerbation)
- The formation of small clusters of immune cells (called granulomas) in parts of your body such as your lymph nodes, eyes, skin, or lungs (sarcoidosis)
- Inflammation of the brain with confusion and fever. This may also include: disorientation, memory problems, seizures (fits), changes in personality and behavior, difficulty speaking, weakness or loss of movement in some parts of your body, and loss of consciousness (encephalitis)
- Inflammation of the spinal cord with pain, numbness, tingling, or weakness in the arms or legs, bladder or bowel problems including needing to urinate more frequently, urinary incontinence, difficulty urinating, and constipation (myelitis)
- Inflammation of the blood vessels (vasculitis)

Additionally, since pembrolizumab was approved in September 2014, the following side effects have been reported by people receiving pembrolizumab.

These side effects were voluntarily reported from a group of people of unknown size. It is not possible to estimate the frequency of these side effects:

- Inflammation of the joints which may include joint pain, stiffness and/or swelling (arthritis)
- Severe responses of the immune system that cause the body to attack its own blood cells, spleen, liver, lymph nodes, skin and brain. This may include fever, rash, inflammation of the liver, yellowing of the skin, an enlarged liver and spleen, low blood counts, and enlarged lymph nodes. The nervous system may also be affected and cause confusion, seizures, and even coma (hemophagocytic lymphohistiocytosis)

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

• Changes in eyesight, eye pain, whitish patches on the skin and hearing loss (Vogt-Koyanagi-Harada syndrome)

• Inflammation and scarring of the bile ducts (tubes that carry digestive fluid that is made in the liver). This can cause symptoms similar to those seen with inflammation of the liver (hepatitis) such as pain in right side of your belly, yellow eyes and skin, feeling tired, and itching (sclerosing cholangitis).

In addition to the above, if you have had an allogeneic stem cell transplant (a procedure in which a person receives blood-forming stem cells from a donor), you may experience graft versus host disease (GvHD), which may include diarrhea, skin rashes, and liver damage, after receiving pembrolizumab. Sometimes this condition can lead to death.

If you have had a solid organ transplant (for example, if you have received a kidney or heart transplant), you may experience rejection of the transplanted organ. Your doctor will monitor you and should tell you what signs and symptoms you should report depending on the type of organ transplant that you have had.

# Potential Risk or Discomfort from Research Procedures

# **Biopsies**

Risks associated with biopsies include pain, redness, swelling, low blood pressure, excessive bleeding, bruising, or draining at the needle site, abnormal wound healing, fever, infection, and allergic reaction to the medication used to numb the skin over the biopsy site. Two to 3% of patients require hospitalization after a tumor biopsy. Rarely, an infection can occur.

#### Magnetic Resonance Imaging (MRI)

If you take part in this research, you will have an MRI (magnetic resonance imaging and/or magnetic resonance spectroscopy). MRI uses a magnet and radio waves to make images (pictures) of the inside of the head and/or body. There have been no ill effects reported from exposure to the magnetism or radio waves used for these studies; however, it is possible that harmful effects could be recognized in the future. A known risk is that the magnet could attract certain kinds of metal that may cause injury to you. We will ask you about metal within your body (this includes certain dyes used in tattoos and body piercings). If there is any question about potentially hazardous metal within your body, you will not be able to participate in this research study. We will also keep the MRI room locked so that no one carrying metal objects enters the room while you are having this scan performed. In addition, the MRI scanner makes a loud buzzing noise that could affect hearing ability. You will be provided with earplugs and assistance

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

in their use in order to protect your hearing. You will be able to communicate with the scanner technologist using an intercom and/or signaling device. The technologist will try to help you feel as comfortable as possible in the scanner. You can ask to stop the scan and be removed from the scanner at any time by using the intercom or signaling device.

There is a very slight risk of an allergic reaction if contrast material is injected. Such reactions usually are mild and easily controlled by medication. If you experience allergic symptoms, a radiologist or other physician will be available for immediate assistance.

**Gadolinium-based** contrast agents (dyes) may increase the risk of a rare but serious disease called nephrogenic systemic fibrosis in people with poor kidney function. Nephrogenic systemic fibrosis triggers thickening of the skin, organs and other tissues. There is no effective treatment for this debilitating disease.

Reproductive risks: You should not get pregnant, breastfeed, or father a baby while in this study. The CNP used in this study could be very damaging to an unborn baby. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), effective May 21, 2010, generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this Federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

What possible benefits can I expect from taking part in this study?

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

We cannot know if you will have any benefit as a result of your participation in the study; it is possible the study treatment may improve your cancer, which may give you relief from some symptoms, improve your quality of life or prolong your survival. However, it is possible that your condition could worsen. Your participation in this study will help to obtain information about treating subjects with CNP.

# Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available
- If you do not follow the study requirements
- If the study is stopped by the sponsor, Institutional Review Board (IRB) or FDA.

# What are my rights in this study?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

# What are the costs of taking part in this study?

Your involvement in this research study is voluntary and you will not be paid for your participation.

The study agent, Pembrolizumab, will be provided free of charge by Merck, Inc. while you are participating in this study. Neither you nor your insurance provider will be responsible for the costs of any research-only tests or procedures. The blood work for research purposes will not be charged to you. It will be paid for by the research study.

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

You and/or your health plan/insurance company will need to pay for some or all of the costs of treating your cancer in this study (i.e., medical history, review of medications, physical exams, performance status, routine blood tests, pregnancy test, x-rays and/or scans for tumor measurement). Some health plans will not pay these costs for people taking part in studies. Check with your health plan or insurance company to find out what they will pay for. Taking part in this study may or may not cost your insurance company more than the cost of getting regular cancer treatment.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at http://www.cancer.gov/clinicaltrials/learningabout.

# Notice for Managed Care (Medicare Advantage Plan) Beneficiaries

Certain services that are required for your care as a participant in a clinical trial can be billed to, and paid by, your medical insurance. These services are referred to as "covered" clinical trial services. However, if you have a Medicare Advantage Plan as part of your medical insurance, this insurance cannot be billed for covered clinical trial services. Instead, traditional Medicare will be billed, and will pay for those services. This has an impact to you. When traditional Medicare pays for such services, you will be responsible for paying the coinsurance amounts applicable to these services, in addition to any other deductibles or co-insurance you may have on your other health coverage. Please speak with a financial counselor to understand what the specific financial impact will be for you associated with participating in this clinical trial.

# What happens if I am injured or hurt because I took part in this study?

If you believe that you are injured as a result of the research procedures being performed, please immediately contact the study doctor.

If injury occurs as a result of your involvement in this research, medical treatment is available from University Hospital, Cleveland Clinic or another medical facility but you/your medical insurance will be responsible for the cost of this treatment. A research injury is an injury that happens as a result of taking part in this research study. If you are injured by a medical treatment or procedure that you would have received even if you weren't in the study, that is not considered a "research injury". There are no plans for payment of medical expenses or other payments, including lost wages, for any research related injury. To help avoid injury, it is very important to follow all study directions.

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

Further information about research-related injuries is available by contacting the Cleveland Clinic Institutional Review Board at (216) 444-2924 or University Hospitals Cleveland Medical Center's Research Subject Rights phone line at (216) 983-4979.

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

# ADDITIONAL STUDIES SECTION: Additional Research Biopsy

# This section is about optional studies you can choose to take part in:

This part of the consent form is about optional studies that you can choose to take part in. You will not get health benefits from any of these studies. The researchers leading this optional study hope the results will help other people with cancer in the future.

The results will be added to your medical records and you or your study doctor will know the results.

You will not be billed for this optional study. You can still take part in the main study even if you say "no" to this additional optional study. If you sign up for but cannot complete any of the studies for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for each of the following studies.

# **Optional Research Biopsy – post treatment**

If you choose to take part in this study, you will have an additional research biopsy.

If you agree to have this additional research biopsy it would involve the removal of a small (pencil eraser-sized) circle of tumor using a cookie cutter-like instrument. The duration of the biopsy procedure is approximately 30 minutes. The biopsy instrument will be placed into the tumor by a physician. The procedure will be done using local anesthesia to minimize discomfort from the biopsy. During a biopsy of the breast, you will be asked to lie flat and a doctor will clean the area on your breast. The doctor will then numb the area with a local anesthetic so that you do not feel the biopsy. The doctor will ask you to hold your breath and not move while he or she places the needle into your tumor and withdraws a small core of tissue which remains trapped inside the needle. This tissue sample will then be forwarded to a research laboratory for further studies. This will help the researchers understand the differences before your treatment on the main research study, and after your treatment on the main research study.

| I agree to undergo an additional research biopsy after main study treatment: | | |
|---|---|---|
| Yes | No | Initials |
| CASE 6115 | | |

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

# HIPAA AUTHORIZATION

Authorization to Use or Disclose (Release) Health Information that Identifies You for a Research Study

If you volunteer to participate in this research, your protected health information (PHI) that identifies you will be used or disclosed to Joseph Baar MD, and the research study staff at Cleveland Clinic and/or University Hospitals for the purposes of this research and to Case Western Reserve University for administration.

The PHI that we may use or disclose (release) for this research may include your name, address, phone number, date of birth, Social Security number, information from your medical record, lab tests, or certain information relating to your health or condition..

Some of the tests and procedures done solely for this research study may also be placed in your medical record so other doctors know you are in this study. Upon completion of the study, you may have access to the research information that is contained in your medical record.

In addition to the investigators and research staff listed above, your PHI may be looked at by other groups involved with the study such as the Cleveland Clinic Institutional Review Board, the University Hospitals Institutional Review Board and the Case Comprehensive Cancer Center Protocol Review and Monitoring Committee. Your PHI may also be used by and/or disclosed (released) to:

- Merck Pharmaceuticals, and its study monitors and representatives
- Case Comprehensive Cancer Center members and collaborators
- The Food and Drug Administration;
- The Department of Health and Human Services;
- The National Cancer Institute (NCI);
- Other Institutional Review Boards:
- Data Safety and Monitoring Boards;

Once your personal health information is released it may be re-disclosed and no longer protected by privacy laws.

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

Your research information may be used and disclosed indefinitely, but you may stop these uses and disclosures at any time by writing to:

Joseph Baar, MD or Case Comprehensive Cancer Center University Hospitals Cleveland Medical Center 11100 Euclid Ave. Cleveland, OH 44106 Jame Abraham, MD
Case Comprehensive Cancer Center
Cleveland Clinic
9500 Euclid Ave.
Cleveland, OH 44195

Your participation in the research will stop, but any information previously recorded about you cannot be removed from the records and will continue to be used as part of this research. Also, information already disclosed outside the Cleveland Clinic and/or University Hospitals cannot be retrieved. This will not affect your rights to treatment or benefits outside the research study.

The Cleveland Clinic and/or University Hospitals will not use your information collected in this study for another research purpose without your written permission; unless the Cleveland Clinic Institutional Review Board (IRB) and/or University Hospitals Institutional Review Board assures your privacy and confidentiality is protected. The IRB is a committee whose job it is to protect the safety and welfare of research subjects.

By signing this informed consent form, you are authorizing such access to your research and medical record information. If you choose not to sign this consent form, you will not be able to participate in this research study. This Authorization does not have an expiration date.

# Voluntary Participation

Your participation in this research study is voluntary. Choosing not to participate will not alter your usual health care or involve any penalty or loss of benefits to which you are otherwise entitled. If you decide to join the study, you may withdraw at any time and for any reason without penalty or loss of benefits. If information generated from this study is published or presented, your identity will not be revealed.

In the event new information becomes available that may affect the risks or benefits associated with this study or your willingness to participate in it, you will be notified so that you can decide whether or not to continue participating.

# Questions about the Research

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

Project Title: CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

If you have any questions, you can ask the Principal Investigator and/or research staff at 216-844-8571.

### Emergency or after-hours contact information

If you are a University Hospitals patient, and you need to contact study staff outside normal business hours, you may contact 216-844-3951 and you will be transferred to the answering service, which can put you in contact with Dr. Baar or the oncologist (cancer doctor) on call.

If you are a Cleveland Clinic patient, you should contact the page operator at (216) 444-2200 or toll free at (800) 223-2273, and ask for the oncologist (cancer doctor) that is on call.

# Where Can I Get More Information?

If the researchers cannot be reached, or if you would like to talk to someone other than the researcher(s) about: concerns regarding the study, research participant's rights; research-related injury; or other human subjects issues, you may contact the Institutional Review Board (IRB) at Cleveland Clinic IRB 216-444-2924 or the University Hospitals Cleveland Medical Center's Research Subjects Rights Phone line at 216-983-4979.

You may call the National Cancer Institute's Cancer Information Service at: 1-800-4-CANCER (1-800-422-6237)

You may also visit the NCI Web site at http://cancer.gov/

- For NCI's clinical trials information, go to: http://cancer.gov/clinicaltrials/
- For NCI's general information about cancer, go to http://cancer.gov/cancerinfo/

You will get a copy of this form. If you want more information about this study, ask your study doctor.

# **US National Institutes of Health (NIH) Clinical Trial Database:**

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, if applicable, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

CASE 6115

Protocol version date: 05.31.21 Consent version date: 03.15.2022

IRB APPROVAL DATE: 3/23/2022 IRB EFFECTIVE DATE: 3/23/2022 IRB EXPIRATION DATE: 6/23/2022

#### CONSENT FOR CANCER RESEARCH

**Project Title:** CASE 6115 Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for

Metastatic Triple-Negative Breast Cancer **Sponsor:** Case Comprehensive Cancer Center

Principal Investigator(s): Joseph Baar, MD, University Hospitals Cleveland Medical Center

Jame Abraham, MD, Cleveland Clinic

# **Signature**

Signing below indicates that you have been informed about the research study in which you voluntarily agree to participate; that you have asked any questions about the study that you may have; and that the information given to you has permitted you to make a fully informed and free decision about your participation in the study. By signing this consent form, you do not waive any legal rights, and the investigator(s) or sponsor(s) are not relieved of any liability they may have. A copy of this consent form will be provided to you.

| Signature of Participant | Date | Printed Name of Participant |
|---|---|---|
| Signature of Witness | Date | Printed Name of Witness |
| I have discussed the information conta<br>opinion that the participant understand<br>with this research study. | | ent with the participant and it is my, alternatives and procedures involved |
| Signature of Person Obtaining Conser | nt Date | |
| Printed Name of Person Obtaining Co | onsent | |

**CASE 6115** 

Protocol version date: 05.31.21 Consent version date: 03.15.2022